CLINICAL TRIAL: NCT01706068
Title: Transient ECG Changes in Patients With Acute Biliary Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Inna Rozenfeld , MD, Principal Investigator, Ziv Hospital
Other Study IDs: ECGCTIL
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Acute Cholecystitis; Biliary Colic; Acute Cholangitis
Keywords: acute ECG changes; acute illness of gallbladder; acute illness of biliary tract
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background:

The importance of ischemic ECG changes including St segment elevation, ST segment depression or T wave inversion that indicate myocardial ischemia are well established and require appropriate investigation and treatment.

However, there is an abundance of clinical situation, with apparently ischemic ECG change not indicate traditionally coronary artery related ischemia and therefore require prompt recognition and treatment of underlying condition, that may be serious and life-threatened. For example of such conditions are pericarditis, myocarditis, aortic dissection, electrolyte abnormalities, intracranial hemorrhage and hypothermia.

Together with them, an ECG ST segment changes may appeared in abdominal serious illness such as pancreatitis and cholecystitis(17,18,19,20,23). Whereas in pancreatitis various vasoactive and toxic for myocardium substances released, the cause of ST segment changes in cholecystitis are discussed and includes tachycardia , vagal reflexes, changed in plasma rennin activity resulted by distension of the gallbladder.

The certain proportion of the patients with ECG changes actually didn't have coronary artery disease(9,15) or other acute cardiac condition and therefore require treatment of the underlie illness only without spend the time for cardiac investigation or special treatment(1,3,4,7,8). Some kind of treatment may be even harmful for the patients with abdominal illness such as thrombolytic, anticoagulant, aggressive antiaggregant therapy or unnecessary cardiac catheterization.

In the medical literature the investigators found some case reports and works about the ECG changes in acute biliary disease in patient with knowing cardiac disease and without it, but actually incidence of ECG changes that suggest but not represent an acute coronary illness isn't knowing.

Therefore this is necessary to investigate actually incidence of ECG changes that mimic acute coronary syndrome in acute cholecystitis and acute biliary disease and determined clinical and laboratory characteristics that helps to differentiate this patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from age 18 and up to 75years old.
2. Causes of admission to the ED are acute cholecystitis, biliary colic, acute cholangitis
3. The patient is willing to participate in the study and is able to sign an informed consent form.

Exclusion Criteria:

1. Elective hospitalization with known and not acute condition.
2. Inability to give inform consent .
3. Sepsis as complication of illness.
4. Chronic ECG changes known by medical history.
5. Knowing history of IHD.
6. Previous cardiac catheterization with documented stenosis of at least 1 major coronary artery equal or more 50%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ECG changes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2014-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel